CLINICAL TRIAL: NCT05475639
Title: Axillary Phonophoresis Versus Post Isometric Facilitation in the Treatment of Shoulder Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Abdel Basset Ali Elsayed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003719
Record Dates: First submitted 2022-07-20; First posted 2022-07-27 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: adhesive capsulitis; post isometric facilitation; axillary phonophoresis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: this trial has three group; two experimental and one control
Who Masked: Participant
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- axillary diclophenac phonophoresis ( diclophen gel "voltaren gel") (Experimental): the subject in the axillary diclophenac phonophoresis group will receive axillary diclophenac phonophoresis using ultrasound 1 MHz to increases the absorbtion. Diclofenac phonophoresis will be applied beside conventional therapy program ,Apply the diclophen gel (voltaren gel) on the head of the US in the axillary pouch of the capsule at 1.5 W\cm2 for 10 minutes as pulsed U.S. the group will be treated for 4weeks, 3 sessions per week and all patients will be assessed pre and post intervention.
  Interventions: Other: Axillary Diclofenac phonophoresis
- Post isometric Facilitation Techniques. (Experimental): the subject in the Post isometric Facilitation Techniques group will be treated by applying isometric contraction followed by isometric relaxation followed by stretching to the target muscle .when performing isometric facilitation with the shoulder in flexion , the patient was seated with his\her back supported and the therapist standing facing the patient's painful shoulder .the patient's shoulder joint was flexed to the maximum available range with the elbow completely flexed .the patient performed isometric contraction of the shoulder extensors against maximum resistance provided by the therapist .this contraction will last for 10 seconds followed by relaxation for 5 seconds .this contraction will allow the shortened shoulder extensors to relax and permit easier stretching.the group will be treated for 4weeks, 3 sessions per week and all patients will be assessed pre and post intervention.
  Interventions: Other: Post isometric facilitation
- traditional physiotherapy (infrared, supervised exercise program, home exercise program) (Active Comparator): The traditional physical therapy program, which includes Infrared (IR) lambs apply heat to deep joints such as shoulder joint. Avoid deltoid muscle; apply over thin, bony areas for maximum penetration.
  supervised exercise program are self-exercise included: 1-Codmans or pendulum exercise (circumduction): It should be done 5 times daily in 5 to 10 minute sessions Passive stretching exercise (for shoulder extensors, abductors, and internal rotator) home exercise program includes the same exercise as in supervised exercise program. The participant will instruct to perform exercises1-2 times/day within pain -free ROM.
  the group will be 4weeks, 3 sessions per week and all patients will be assessed pre and post intervention.
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Other: Axillary Diclofenac phonophoresis — axillary diclophenac phonophoresis (voltaren gel) will be received three times per week for four weeks
  Arms: axillary diclophenac phonophoresis ( diclophen gel "voltaren gel")
Other: Post isometric facilitation — Post isometric facilitation exercise will be received three times per week for four weeks
  Arms: Post isometric Facilitation Techniques.
Other: Traditional physiotherapy — Traditional physiotherapy will be received three times per week for four weeks
  Arms: traditional physiotherapy (infrared, supervised exercise program, home exercise program)

SUMMARY:
the aim of this study is to compare the effect of Axillary Phonophoresis versus Post isometric facilitation in subjects with Adhesive capsulitis

DETAILED DESCRIPTION:
Adhesive Capsulitis is a common cause of shoulder pain and disability and also a condition involving glen humeral pain and loss of motion. It is characterized by significant restriction of both active and passive motion that occurs in the absence of a known intrinsic shoulder disorder. The intervention strategies for AC include a trial of conservative therapy followed by more invasive procedures.it may be primary-onset is generally idiopathic or Secondary- results from known cause. Clinically, patients may present with pain and mild restriction of movement which can lead to a gross loss of function predisposing factor or surgical event . it is most frequent in women, diabetic population and patient older than 40 years .It is described as having 3 stages. Stage Ⅰ involves pain (freezing or painful stage) and lasts from 3 to 9 months and is characterized by an acute synovitis of the glen humeral joint. Stage Ⅱ (frozen or transitional stage) includes pain and restricted movement and lasts from 4 to 12 months. Stage Ⅲ (thawing stage) involves painless restriction and lasts from 12 to 42 months. Contributing factors include diabetes mellitus, stroke, thyroid disorder, dupuytren disease, complex regional pain syndrome and metabolic syndrome.

Axillary Phonophoresis and Post isometric facilitation play a major role in the treatment of adhesive capsulitis so this trial was conducted to determine which one has superiority. this trial has three groups. two experimental and one control group. pain ,function, pressure pain threshold will be measured.

ELIGIBILITY:
Inclusion Criteria:

* The patient age will range from 30to 40years old from both sexes (male and female).
* All recruited subjects in the 2nd stage of adhesive capsulitis (transitional stage).
* The patient will be diagnosed and referred by orthopedist as Adhesive capsulitis.
* The diagnosis will be confirmed by shoulder MRI.
* The diagnosis will be confirmed by shrug test.
* The patient will be referred by anterior shoulder pain or anterolateral shoulder pain.
* Inclusion requirement include two or more of the following pain complaints: Grooming ones hair, Scratching your back and getting dressed, Overhead activities or Difficulty in the action of throwing the ball and giving a high -five.
* All patients will sign the informed consent before joining the study.

Exclusion Criteria:

* Previous fracture with or without internal fixation in the shoulder joint
* Any previous surgery in the shoulder joint and patient with tendon calcification
* Local corticosteroid injection to the affected shoulder within the last three months or recent ones (Michener et al, 2004).
* Neuromuscular disease
* Rotator cuff tear
* History of metastatic cancer or diagnosis of cancer within 12 months
* Unstable angina

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-25 (Estimated); Primary Completion 2023-06-05 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to six weeks
  numerical rating scale (NRS) will be used for assessment of pain intensity. the scale from 0 to 10 where 0 is no pain and 10 is the worst pain
pressure pain threshold | up to six weeks
  commander algometer will be used for measuring pressure pain threshold
shoulder range of motion | up to six weeks
  digital goniometer will be used for measuring range of motion
shoulder functional activity | up to six months
  Disability of the Arm, Shoulder, and Hand questionnaire (DASH) will be used for measuring shoulder function activity. it is a shortened version of the DASH questionnaire that uses 11 items to measure the degree of difficulty in performing various physical activities due to a shoulder, arm, or hand problem (6 items); the severity of pain and tingling (2 items); and the problem's effect on social activities, work, and sleep (3 items)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa El-sayed, Bachlore, Principal Investigator — Cairo University